CLINICAL TRIAL: NCT03107702
Title: Relationship Between Melatonin Level and Postoperative Analgesia Consumption in Bariatric Surgery Patients.
Brief Title: Melatonin Level and Postoperative Analgesia Consumption in Bariatric Surgery Patients.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Mehmet Ali Erdoğan, Associate professor, Inonu University
Other Study IDs: MAE5
Record Dates: First submitted 2017-03-29; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Bariatric Surgery; Melatonin; POSTOPERATIVE PAIN
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Melatonin and bariatric surgery: the relationship between melatonin level and analgesia requirement.
  Interventions: Diagnostic Test: melatonin

INTERVENTIONS:
Diagnostic Test: melatonin — the relationship between melatonin level and analgesia requirement.

SUMMARY:
Bariatric surgical procedures are associated with low short-term mortality and may be associated with long-term reductions in all-cause, cardiovascular, and cancer-related mortality. This surgeries are major surgeries include risk of mortality still.

Melatonin is a hormone secreted from the pineal gland. Melatonin is an antioxidant, antinociceptive, hypnotic, anticonvulsant, neuroprotective, anxiolytic, sedative and analgesic. Melatonin is neurohormone with the profile of a novel hypnotic-anesthetic agent.

The purpose of this study is to investigate the preoperative, perioperative and postoperative melatonin levels in bariatric surgery under general anesthesia and to investigate the relationship between melatonin level and analgesia requirement.

DETAILED DESCRIPTION:
Bariatric surgical procedures are associated with low short-term mortality and may be associated with long-term reductions in all-cause, cardiovascular, and cancer-related mortality. This surgeries are major surgeries include risk of mortality still.

Melatonin is a hormone secreted from the pineal gland. Melatonin is an antioxidant, antinociceptive, hypnotic, anticonvulsant, neuroprotective, anxiolytic, sedative and analgesic. Irregularity of melatonin secretion causes a sleep irregularities, psychosis in intensive care unit and some behavioral disorder. The hypnotic, antinociceptive, and anticonvulsant properties of melatonin endow this neurohormone with the profile of a novel hypnotic-anesthetic agent.

The purpose of this study is to investigate the preoperative, perioperative and postoperative melatonin levels in bariatric surgery under general anesthesia and to investigate the relationship between melatonin level and analgesia requirement.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) 3-4 status, aged between 18-65 years who are scheduled to undergo bariatric surgery.

Exclusion Criteria:

Patients with cardiovascular and pulmonary disease, those with ASA III-IV and propofol, fentanyl, remifentanil and rocuronium allergy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients of American Society of Anesthesiologists (ASA) 1-2 status, aged between 18-65 years who are scheduled to undergo bariatric surgery.
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2017-03-29 (Actual); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-07-30 (Estimated)

PRIMARY OUTCOMES:
Melatonin Level | Change from Baseline melatonin at postoperative 24 hours
  Melatonin is a hormone secreted from the pineal gland. It shows a daily biorhythm. Melatonin level can be measured in the blood and in urine collected for 24 hours.

SECONDARY OUTCOMES:
Morphine consumption | change from postoperative up to 24 hours
  Morphine is analgesic agent. It will used postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Türkan Toğal, Prof., Study Director — Inonu University Faculty of Medicine
Locations (1):
- Inonu university, Malatya, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naguib M, Gottumukkala V, Goldstein PA. Melatonin and anesthesia: a clinical perspective. J Pineal Res. 2007 Jan;42(1):12-21. doi: 10.1111/j.1600-079X.2006.00384.x. PMID 17198534
- [Background] Gogenur I, Ocak U, Altunpinar O, Middleton B, Skene DJ, Rosenberg J. Disturbances in melatonin, cortisol and core body temperature rhythms after major surgery. World J Surg. 2007 Feb;31(2):290-8. doi: 10.1007/s00268-006-0256-5. PMID 17180564
- [Background] Hansen MV. Chronobiology, cognitive function and depressive symptoms in surgical patients. Dan Med J. 2014 Sep;61(9):B4914. PMID 25186550
- [Derived] Altunkaya N, Erdogan MA, Ozgul U, Sanli M, Ucar M, Ozhan O, Sumer F, Erdogan S, Colak C, Durmus M. Changes in Melatonin, Cortisol, and Body Temperature, and the Relationship Between Endogenous Melatonin Levels and Analgesia Consumption in Patients Undergoing Bariatric Surgery. Obes Surg. 2018 Oct;28(10):3186-3192. doi: 10.1007/s11695-018-3313-x. PMID 29785473